CLINICAL TRIAL: NCT02530892
Title: Measuring the Relationship Between Ooocyte and Embryo Mechanical Properties and Embryo Development After In Vitro Fertilization
Brief Title: Correlation Between Oocyte and Embryo Mechanical Properties on Embryo Development and Clinical Pregnancy After In Vitro Fertilization
Acronym: EMECH
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: 31948
Record Dates: First submitted 2015-08-04; First posted 2015-08-21 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Infertility; Pregnancy, Multiple
Keywords: embryo; in vitro fertilization; IVF
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Measurement Group: This group contains oocytes and embryos which have their mechanical properties (elasticity and viscosity) measured prior to fertilization (oocytes) or within 24 hours after fertilization (embryos). The investigators are calling this mechanical measurement the "EmbryoHug." All participants in the study will have half their embryos measured in this group. Outcomes will be evaluated after 6 days of embryo culture, at the time of pregnancy test, at 5-6 weeks, and at 8-10 weeks, and correlated with EmbryoHug parameters.
  Interventions: Procedure: EmbryoHug

INTERVENTIONS:
Procedure: EmbryoHug — An oocyte or embryo will be gently held by a micropipette, and a small inward pressure will be applied to the edge of the oocyte or embryo. The response of the embryo to this pulling force will allow the investigators to measure its stiffness and viscosity. The term "micropipette aspiration" refers to the pressure applied to the edge of the embryo -- this procedure is not invasive and does not involve any sort of puncture or removal of material from the oocyte or embryo.
  Other Names: Micropipette Aspiration; Mechanical Measurement

SUMMARY:
The purpose of this study is to determine whether oocyte and embryo mechanical properties measured during in vitro fertilization can predict embryo development outcomes and clinical pregnancy.

DETAILED DESCRIPTION:
In the current practice of in vitro fertilization (IVF), clinicians often transfer multiple embryos to the patient at once in an effort to maximize chances of pregnancy. This practice results in a high rate of multiple births which increase the risks of complications for mothers and children.

The investigators in this study have developed a novel, noninvasive marker of embryo viability which is based on measuring embryo mechanical properties at the oocyte or the 1-cell stage. The investigators would like to test whether human oocyte or embryo mechanical properties are predictive of subsequent development, clinical pregnancy, and compare their predictive power to that of a morphological assessment (the current gold standard). Using this approach, clinicians could more confidently move toward single embryo transfer, provided more individualized counseling for patients undergoing oocyte cryopreservation, as well as improve pregnancy rates after IVF.

This is a pilot observational study. Although investigators will measure the mechanical properties of all participant oocytes and embryos, no prediction of embryo viability will be made, and there will be no intervention in choosing which embryos to transfer to participants. The data from this study will eventually be used to find a range of oocyte and embryo mechanical parameters which are predictive of high developmental potential, and will serve as the basis for an interventional study in the future.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 21 and 45
* Undergoing intra-cytoplasmic sperm injection (ICSI) at Stanford Fertility, Shenzhen IVF clinic, or Taiwan IVF group between August 2015 and August 2018

Exclusion Criteria:

* Using gestational carrier or donor eggs
* Using cryopreserved eggs
* Fewer than 5 oocytes collected

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients undergoing in vitro fertilization at the Stanford IVF clinic, the Shenzhen IVF clinic, or Taiwan IVF group are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2015-08; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy (8-10 weeks) | 8-10 weeks
  Positive result is determined by presence of intrauterine gestational sac and fetal heartbeat. Outcome will record number of gestational sacs with heartbeat present.

SECONDARY OUTCOMES:
Blastocyst grade (Gardner scale) | 5-6 days
  If the embryo reaches the blastocyst stage, its inner cell mass and trophectoderm will be graded according to Gardner's criteria. If no blastocyst is formed, that will be recorded as well.
Pregnancy test result (based on human chorionic gonadotropin (hCG) levels) | 2-3 weeks
  Outcome will be recorded as either positive or negative.
Clinical pregnancy (5-6 weeks) | 5-6 weeks
  Positive result is determined by presence of intrauterine gestational sac and fetal heartbeat (although sometimes the heartbeat does not show up for another week or two). Outcome will record number of gestational sacs.
Fertilization rate | 1 day
  For oocytes measured, the fertilization of oocytes will be recorded.
Day 3 morphology | 3 days
  For oocytes measured, the day 3 morphology of embryos will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Baker, MD, Principal Investigator — Stanford University
Locations (3):
- Stanford University IVF clinic, Stanford, California, United States
- Shenzhen Army and Police Hospital--Reproductive Unit, Shenzhen, China
- Taiwan IVF Group, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Upon publication of study results, we may include de-identified participant data for people who wish to conduct their own analysis.